CLINICAL TRIAL: NCT03042208
Title: Ripple Effect of a Nationally Available Weight Loss Program on Untreated Family Members
Brief Title: Weight Watchers and Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-260
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to Weight Watchers in-person meetings and online tools.
  Interventions: Behavioral: Weight Watchers
- Self-Guided Control Group (Other): Received handout with basic weight management advice.
  Interventions: Other: Self guided handout

INTERVENTIONS:
Other: Self guided handout — Written handout with basic weight management strategies
  Arms: Self-Guided Control Group
Behavioral: Weight Watchers — Access to Weight Watchers in-person meetings and online tools
  Arms: Intervention

SUMMARY:
Research suggests that when one spouse loses weight, the other spouse does too. This study will examine whether a ripple effect is observed in untreated spouses and children of individuals participating in a nationally available weight loss program. Participants will be randomly assigned to either receive Weight Watchers immediately or at the end of a 6-month waiting period. Participants and untreated spouses (and any children in the home) will be assessed at baseline, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 27.0-40.0 kg/m2
* married or living with a significant other who had a BMI > 25 kg/m2

Exclusion Criteria:

* currently in a weight loss program, dieting, or taking medications that might affect weight
* had participated in a weight loss program in the past year
* lost > 5% of their body weight in the past 6 months
* were planning to or had undergone weight loss surgery
* had any orthopedic limitations or contraindications to physical activity
* were pregnant, lactating, or less than 6 months postpartum, or were planning to become pregnant in the next year
* reported uncontrolled hypertension, history of coronary heart disease, stroke, or peripheral arterial disease; reported chronic gastrointestinal disease
* endorsed having hepatitis B or C, cirrhosis, or HIV
* had a history of cancer within the past 5 years
* reported a significant psychiatric illness that might interfere with completion of the study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 0, 3, and 6 months
  body weight measured in kg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McManus-Shipp KE, Cornelius T, Wojtanowski AC, Leahey T, Foster GD, Gorin AA. Family functioning and the implications for adult weight management. Fam Syst Health. 2025 Mar;43(1):157-161. doi: 10.1037/fsh0000929. Epub 2024 Sep 16. PMID 39283252
- [Derived] Gorin AA, Lenz EM, Cornelius T, Huedo-Medina T, Wojtanowski AC, Foster GD. Randomized Controlled Trial Examining the Ripple Effect of a Nationally Available Weight Management Program on Untreated Spouses. Obesity (Silver Spring). 2018 Mar;26(3):499-504. doi: 10.1002/oby.22098. Epub 2018 Feb 1. PMID 29388385